CLINICAL TRIAL: NCT07224867
Title: The Effects of Liquid IV's Multi-Ingredient Recovery Supplement, on Muscle Recovery Following Exercise: A Randomized Crossover Study
Brief Title: The Effects of Liquid IV's Multi-Ingredient Recovery Supplement on Muscle Recovery Following Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00089373
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Muscle Damage; Strength Recovery; Perceived Recovery; Perceived Muscle Soreness; Physical Performance; Muscle Recovery
Keywords: muscle damage; muscle recovery; strength recovery; physical performance; perceived recovery; perceived muscle soreness

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, crossover study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proprietary post workout recovery supplement (Experimental): Liquid I.V. post workout recovery powder mixture
  Interventions: Dietary Supplement: proprietary post workout recovery supplement
- Control Treatment (Placebo Comparator): inactive/inert placebo mixture
  Interventions: Dietary Supplement: Control placebo

INTERVENTIONS:
Dietary Supplement: proprietary post workout recovery supplement — proprietary post workout recovery supplement
  Arms: proprietary post workout recovery supplement
Dietary Supplement: Control placebo — inactive/inert placebo mix
  Arms: Control Treatment

SUMMARY:
The purpose of this study is to evaluate the efficacy of a multi-ingredient recovery supplement . The research will focus on strength recovery and performance maintenance assessing reductions in soreness and inflammation, as well as muscle repair and damage mitigation. By investigating these key recovery metrics, this study aims to investigate the efficacy of this supplement as a solution for active individuals seeking to optimize post-exercise recovery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18-55 years old.
* Must be recreationally trained or trained/developmental as previously defined (McKay et al., 2021).
* Able to read and write in English.
* Cessation of current use of tart cherry extract, protein powders, essential amino acids/BCAAs, collagen/collagen peptides, or anabolic agents for a minimum of 1-weeks prior to, and throughout the duration of the study.
* Willing to maintain regular supplement routine otherwise during the trial, and will not introduce or discontinue a supplement, other than what was previously mentioned.
* Will not participate in any strenuous exercise for a minimum of 1-week prior exercise performance assessments, as well as during the days of exercise testing. Strenuous exercise as defined for this study includes ½ and full marathons (or more), heavy (i.e.,>80% 1RM) lifting, and any high intensity, physical activity that could make your muscles sore.
* During the study, you agree not to take any NSAIDs or other anti-inflammatory medications.

Exclusion Criteria:

* Sedentary
* Vegan, unwilling to consume animal bovine collagen
* Highly trained/national level or professional athlete
* Known diagnosis of any cardiovascular, metabolic, musculoskeletal, endocrine, or renal disease/disorder.
* Recent musculoskeletal injury (<3-months)
* Recent orthopaedic surgery (<12-months)
* History or current malignancy.
* Current respiratory infection (i.e., cold) or high temperature (fever) within the past 4-weeks.
* Previous gastrointestinal surgery within the past 12 months.
* Regular smoker.
* Regular drinker (>14 drinks per week).
* Those regularly using anti-inflammatory drugs within the last 4-weeks.
* Current use of prescription medications that may influence adaptation to exercise (hormone therapies, peptides, etc.).
* Allergies to study-related materials.
* Any condition that impairs their ability to complete the required exercises.
* Female subjects must not be pregnant or lactating.
* Are unable to provide informed consent or are non-English speakers.
* Presently using GLP-1 medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Lower Body Power and Force Generation (Maximal Countermovement Jump (CMJ)) | Taken at baseline testing, 24hr, 48hr, and 72hr.
  The force plate platform consists of two force plates (left & right) containing four force sensors which measure ground reaction force. The sensors are connected to a laptop and analyzed using Mechanography GRFP Research Edition® software (version 4.2-b05.53-RES).
  Subjects will perform three maximal vertical CMJs on a calibrated force plate. Subjects will be instructed to stand upright on the center of the force plate with feet shoulder-width apart and hands placed on the hips. Subjects will perform a maximal effort vertical jump with proper form and instructed to land with soft knees and remain still after each jump for data capture. A 30sec rest period will be provided between each trial. Data will be used to assess maximum force output (Fmax), rate of force development (RFD), jump height (inches), and maximum power (Pmax). Force curves will be reviewed for each trial, and results averaged. This will quantify full-body mechanical power under standardized, reproducible conditions.
Lower-Body Strength (Biodex Dynamometry) | Tested at baseline, 24hr, 48hr, and 72hr.
  Participants will complete isometric and isokinetic strength assessments, unilaterally on the dominant leg, of knee extension (ext) and flexion (flx) using a Biodex System 4 Pro dynamometer (Biodex Medical Systems, Shirley, NY). Proper positioning and stabilization will be ensured per manufacturer guidelines.
  Isometric testing - knee joint will be fixed @60° of flexion. Participants will perform 3 maximal effort ext/flx contractions, each lasting 5sec, with 5sec of rest between efforts. Highest recorded torque value across the 3 trials will be analyzed.
  Subjects will then complete isokinetic testing consisting of 5 maximal concentric knee ext and flx at an angular velocity of 60°/s. Full range of motion will be established prior to testing. Peak torque and average torque across all 5 repetitions will be recorded for analysis.
  All torque values will be gravity-corrected by the system software, and same technician will conduct all tests for consistency.
Perceived Recovery Status (PRS) Likert Scale | Taken at baseline testing, 24hr, 48hr, and 72hr timepoints.
  The PRS is a composite scale directly proportional to recovery (Laurent, et al. 2011). Hence, the purpose of the scale will be to assess the participant's recovery from the previous exercise session. Subjects will be informed that having no soreness and a high feeling of recovery is a 10, while extreme soreness and low feelings of recovery, leading to limited ability to function, is defined by a range of 0-3, adequate recovery, with some ability to function, is defined by a range of 4-7, and good recovery, with the ability to function normally, is defined by a range of 8-10.
Perceived Body Soreness Likert Scale | Taken at baseline testing, 24hr, 48hr, and 72hr timepoints.
  A 7-point likert scale will be used for lower body muscle soreness, after performing 5 air squats. The Likert scale is a validated instrument designed to assess self reported muscle soreness, measured across a 7-point scale. The scale ranges from 0 (no soreness), to 6 (unbearable soreness), and has good validity and reliability (Impellizzeri, F., et al., 2007).

SECONDARY OUTCOMES:
Body Hydration Status (InBody) | taken during baseline testing only - before exercise and again at ~10min post treatment
  Body hydration status will be assessed using multi-frequency bioelectrical impedance analysis (BIA) (InBody 770, InBody Co., Ltd., Seoul, South Korea). The InBody device uses direct segmental multi-frequency impedance (5 kHz to 1 MHz) to estimate water distribution across body compartments. Measurements will include total body water (TBW), extracellular water (ECW), and intracellular water (ICW) to evaluate fluid compartment status. BIA assessments will be conducted under standardized conditions with participants barefoot, standing upright with arms slightly abducted, and heels positioned on the footplate electrodes. Light, non-conductive clothing will be required, and all metal (e.g., jewelry, watches) are removed before testing. To minimize fluid variability, participants will avoid food, drink, and caffeine for at least 8 hours prior to testing. Measurements will be collected pre-supplementation and post-exercise/post supplement as part of the hydration analysis at baseline only.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sikorski, PhD, Principal Investigator — Applied Science and Performance Institute
Locations (1):
- Applied Science & Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skurvydas A, Brazaitis M, Venckunas T, Kamandulis S. Predictive value of strength loss as an indicator of muscle damage across multiple drop jumps. Appl Physiol Nutr Metab. 2011 Jun;36(3):353-60. doi: 10.1139/h11-023. Epub 2011 May 16. PMID 21574783
- [Background] Shimomura Y, Yamamoto Y, Bajotto G, Sato J, Murakami T, Shimomura N, Kobayashi H, Mawatari K. Nutraceutical effects of branched-chain amino acids on skeletal muscle. J Nutr. 2006 Feb;136(2):529S-532S. doi: 10.1093/jn/136.2.529S. PMID 16424141
- [Background] Connolly DA, McHugh MP, Padilla-Zakour OI, Carlson L, Sayers SP. Efficacy of a tart cherry juice blend in preventing the symptoms of muscle damage. Br J Sports Med. 2006 Aug;40(8):679-83; discussion 683. doi: 10.1136/bjsm.2005.025429. Epub 2006 Jun 21. PMID 16790484
- [Background] Blomstrand E, Eliasson J, Karlsson HK, Kohnke R. Branched-chain amino acids activate key enzymes in protein synthesis after physical exercise. J Nutr. 2006 Jan;136(1 Suppl):269S-73S. doi: 10.1093/jn/136.1.269S. PMID 16365096
- [Background] Impellizzeri FM, Maffiuletti NA. Convergent evidence for construct validity of a 7-point likert scale of lower limb muscle soreness. Clin J Sport Med. 2007 Nov;17(6):494-6. doi: 10.1097/JSM.0b013e31815aed57. PMID 17993794
- [Background] Laurent CM, Green JM, Bishop PA, Sjokvist J, Schumacker RE, Richardson MT, Curtner-Smith M. A practical approach to monitoring recovery: development of a perceived recovery status scale. J Strength Cond Res. 2011 Mar;25(3):620-8. doi: 10.1519/JSC.0b013e3181c69ec6. PMID 20581704